CLINICAL TRIAL: NCT06653660
Title: Exposure to Organochlorine Pollutants and Impact on Development in the Peripubertal Age in Guadeloupe
Acronym: TIMOUNPUBERTY
Status: Recruiting | Type: Observational
Sponsor: Centre Hospitalier Universitaire de la Guadeloupe (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Other Study IDs: PAP_RI2_2019/11
Record Dates: First submitted 2023-09-06; First posted 2024-10-22 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Prenatal Exposure; Postnatal Exposure
Keywords: Prenatal Exposure; Postnatal Exposure; Chlordecone; Persistent Organic Pollutants; Endocrine disruptors; Puberty; Development; Guadeloupe; French West Indies
MeSH Terms: interventions — Restraint, Physical; Blood Specimen Collection; Neuropsychological Tests

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- peripubertal children: Children born from a mother whose pregnancy was included in the Timoun cohort (2004 -2007).
  Interventions: Other: Clinical examination

INTERVENTIONS:
Other: Clinical examination — For the aim of the present study, we will follow-up children born alive in the TIMOUN cohort at peripubertal age. Questionnaires will be administered to parents on the child's health and lifestyle. Stature-weight anthropometric and cardio-dynamic measurements of the child will be obtained. Scores on three cognitive tests will be obtained. Furthermore, steroid hormones and chlordecone in the child's peripheral blood will be determined.
  Other Names: Blood collection,; cognitive tests

SUMMARY:
In the context of environmental pollution of the French West Indies by chlordecone and questions about health consequences, monitoring at the peripubertal age of children born alive in the TIMOUN cohort is justified in several respects: - existence of an already established mother-child cohort whose live-born children will reach peripubertal ages during the period 2020-2022; - opportunity to verify hypotheses put forward on the basis of toxicological data acquired in laboratory animals and the hormonal characteristics of chlordecone (endocrine disruptor); - strong societal demand for such research to be carried out because of concerns about the sensitivity of children and adolescents to the effects of environmental xenobiotics, in particular on sexual development and the age of puberty; - recommendation of the Scientific Council Chlordecone Inserm - InVS; specific action of the National Plan Chlordecone IV.

DETAILED DESCRIPTION:
The French West Indies are permanently polluted by chlordecone. It is an organochlorine insecticide used from 1973 to 1993 in Guadeloupe and Martinique to control banana root borers. Its physico-chemical properties give it great stability and are at the origin of its persistence in the environment. Soil, flora and wildlife pollution from chlordecone in the Caribbean was first documented shortly after its introduction in 1973. However, it was not until 1999 that this pollution was extended to waters intended for human consumption and to various local, vegetable and animal, land and aquatic foodstuffs. The population is also affected, as confirmed by impregnation studies, with exposure nowadays occurring mainly through the consumption of contaminated food. The contamination of the French West Indies populations by this insecticide raises many questions about its possible health consequences. In order to assess the effects of chlordecone exposure on child development in Guadeloupian children, a longitudinal and prospective study, the Timoun mother-child cohort, was initiated. Between 2004 and 2007, women in the second trimester of pregnancy who planned to give birth in the public hospitals of Grande-Terre and Basse-Terre (accounting for 70% of all deliveries in Guadeloupe) were invited to participate in the study. Children born to these included women have been enrolled to several follow-ups during the last years (3, 7, 18 months and 7 years of age).

ELIGIBILITY:
Inclusion Criteria:

* Be born to a mother whose pregnancy was included in the Timoun cohort (2004 - 2007) and whose parents agreed to be contacted later.
* Residing in Guadeloupe at the peripubertal age
* Affiliation to a social security scheme
* Agreement to participate in the study and informed consent signed by the minor
* Study participation agreement and informed consent signed by the parents

Exclusion Criteria:

* Refusal to participate in the research

Ages: 16 Years to 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Be born to a mother whose pregnancy was included in the Timoun cohort (2004 - 2007)
Sampling Method: Non-Probability Sample
Enrollment: 650 (Estimated)
Dates: Start 2022-12-19 (Actual); Primary Completion 2026-12-19 (Estimated); Study Completion 2026-12-19 (Estimated)

PRIMARY OUTCOMES:
Scores from cognitive development tests estimating verbal comprehension verbal comprehension, perceptual reasoning and working memory | At the start of the study (inclusion visit)
  : Cognitive tests (25 min for the 3 Wechsler Intelligence Scale for Children V subscales). The Wechsler Intelligence Scale for Children-V is the most scientifically valid intelligence test for children and adolescents. It can be used to determine a child's or teenager's intelligence quotient (IQ), to obtain their complete cognitive profile and the level of the 5 main components of cognitive intelligence

SECONDARY OUTCOMES:
Age at onset of pubertal development (onset of accelerated growth acceleration of growth rate, modeled on growth curves) | At the start of the study (inclusion visit).
  Collect of the age at which children and adolescents begin to develop adult physical characteristics, such as breasts or pubic hair, and become able to procreate.

OTHER OUTCOMES:
Age at established puberty (period for girls, molting for boys) | At the start of the study (inclusion visit) or through study completion, an average of two years, for girls who had their period and boys molted.
  Collect of the age at which girls had their period and boys molted
Plasma concentrations of steroid hormones | At the start of the study (inclusion visit).
  Blood collection for hormonal and organochlorine pollutants dosage.
Blood pressure | At the start of the study (inclusion visit).
  Seated resting blood pressure will be measured using an automatic tensiometer an automatic blood pressure monitor, with two measurements separated by 15 to 30 minutes.
heart rate | At the start of the study (inclusion visit).
  heart ratewill be measured using an automatic tensiometer an automatic blood pressure monitor, with two measurements separated by 15 to 30 minutes.

CONTACTS AND LOCATIONS:
Overall Officials: Gulen AYHAN, Principal Investigator — CHU of Guadeloupe
Locations (1):
- CHU of Guadeloupe, Pointe-à-Pitre, Guadeloupe, Guadeloupe